CLINICAL TRIAL: NCT01708434
Title: Feasibility Study: Evaluation of the Ulthera® System for Lifting and Tightening of the Knees
Brief Title: Feasibility Study: Evaluation of the Ulthera® System for Treatment of the Knees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ULT-115
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2013-06

CONDITIONS: Skin Laxity
Keywords: Skin laxity; Knees
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ulthera® treatment of the knees (Experimental): Bilateral treatment of the knees using the Ulthera® System
  Interventions: Device: Ulthera® System

INTERVENTIONS:
Device: Ulthera® System — Focused ultrasound energy delivered below the surface of the skin
  Other Names: Ultherapy™ treatment

SUMMARY:
Enrolled subjects will receive one bilateral Ulthera® treatment on the knees. Up to 30 subjects will be enrolled. Study photos will be obtained prior to study treatment, immediately following study treatment, and at each post-treatment follow-up visit. Follow-up visits will occur at 90 and 180 days post-treatment.

DETAILED DESCRIPTION:
This pilot study is a prospective, single-center clinical trial of the Ulthera® System for treating skin laxity on the knees. Global Aesthetic Improvement Scale scores and Patient Satisfaction questionnaires will be obtained at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 30 to 65 years.
* Subject in good health.
* Mild to moderate skin laxity around the knees.
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* Excessive subcutaneous fat around the knees.
* Excessive skin laxity around the knees.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Improvement in overall lifting and tightening of knee skin laxity. | 90 and 180 days post-treatment
  Assessed based on Principal Investigator assessment using the Global Aesthetic Improvement Scale.

SECONDARY OUTCOMES:
Overall improvement in skin laxity. | 90 and 180 days post-treatment
  Determined based on a qualitative masked assessment comparing pre-treatment and post-treatment photographs; subjects' assessment based on the Subject Global Aesthetic Improvement Scale; completion of the Patient Satisfaction Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gold, MD, Principal Investigator — Tennessee Clinical Research Center
Locations (1):
- Tennessee Clinical Research Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Gold MH, Sensing W, Biron J. Use of micro-focused ultrasound with visualization to lift and tighten lax knee skin (1.). J Cosmet Laser Ther. 2014 Oct;16(5):225-9. doi: 10.3109/14764172.2014.949273. Epub 2014 Sep 2. PMID 25065380